CLINICAL TRIAL: NCT05302089
Title: The Effect of Rehabilitation Following Non-surgical Management of Displaced Proximal Humerus Fractures: a Randomized Clinical Trial
Brief Title: Rehabilitation Following Displaced Proximal Humerus Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: University of Southern Denmark (Other); University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHF_rehab
Record Dates: First submitted 2022-03-14; First posted 2022-03-31 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Shoulder Fractures
Keywords: Proximal humerus fractures; Proximal humeral fractures; Randomized controlled trial; Shoulder fractures; Non-operative treatment; Rehabilitation
MeSH Terms: conditions — Shoulder Fractures | interventions — Pain Management

STUDY DESIGN:
Masking Description: Patients will not know the direction of our hypothesis. A blinded statistician will perform the primary analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One-time physiotherapy instruction (Experimental): One-time physiotherapy instruction and no usual rehabilitation care
  Interventions: Other: Pain management and shoulder bandage; Other: One-time physiotherapy instruction
- Usual rehabilitation care (Active Comparator): One-time physiotherapy instruction and usual rehabilitation care
  Interventions: Other: Pain management and shoulder bandage; Other: One-time physiotherapy instruction; Other: Usual rehabilitation care

INTERVENTIONS:
Other: Pain management and shoulder bandage — All Patients receive standard pain management according to the local guidelines and a sling and swathe on the day of injury. After 10 to 14 days, all patients will receive a sling for optional use for one to two weeks and be randomized after oral and written informed consent.
Other: One-time physiotherapy instruction — Patients are offered a one-time physiotherapy instruction about the course of pain and suggestions for quick and safe return to activities of daily living within the first three months post-injury.
Other: Usual rehabilitation care — At the visit 10-14 days after the injury, the orthopaedic consultant (senior author SB) will refer the patient to usual rehabilitation care with a physiotherapist in a municipality close to the patient´s home. The physiotherapist then schedules the start date, typically three weeks after the injury. The rehabilitation content and duration is planned according to the choice of the local treating physiotherapist in consultation with the patient.
  Arms: Usual rehabilitation care

SUMMARY:
Proximal humerus fractures (PHFs) are the third most common non-vertebral fractures in the elderly. Most elderly experience loss of function following a PHF regardless of treatment. A Cochrane review from 2015 concluded that surgical management is not superior to non-surgical management, and that the optimal non-surgical management after PHF is not known. Therefore, the aim of this study is to evaluate the effectiveness of usual rehabilitation care after displaced PHF compared with one-time physiotherapy instruction.

DETAILED DESCRIPTION:
Proximal humerus fractures (PHFs) are the closely related to osteoporosis. The lifetime risk of suffering a PHF in females aged 50 or above is 13%. About half of the fractures are minimally displaced and usually managed by short immobilization, analgetics, and early mobilization. The remaining half of the patients suffer from displaced fractures, traditionally managed surgically by open reduction and internal fixation or shoulder replacement. Within the last decades, an increasing number of high-quality randomized controlled trials (RCTs) and meta-analyses have failed to document the superiority of surgical management in displaced PHFs. Therefore, an increasing number of patients are being offered nonsurgical treatment consisting of immobilization followed by rehabilitation that may vary across countries and regions. Most elderly experience loss of function following a PHF regardless of treatment. However, optimal management and recovery of function are paramount to prevent a substantial impact on the patient's independent living and morbidity. A systematic review and metaanalysis from 2021 concluded a need for high-quality RCTs to substantiate the current evidence regarding the need for supervision after a PHF.

It is assumed that rehabilitation delivered as structured training benefits patients with PHFs, but this is not known from current evidence. It is possible that patients are even harmed with intensive training programmes. Most RCTs with a non-surgically treated group use the same exercise intervention in the two groups to best identify the difference between surgery and non-surgical treatment. Therefore, the effect of training cannot be concluded from these studies. This is supported by an expectation of more nonsurgically treated displaced PHFs due to the growing evidence of no benefit from surgery. The current study is a prerequisite for future rehabilitation studies comparing different training modalities. Therefore, this study aims is to evaluate the effectiveness of usual rehabilitation care after displaced PHF compared with one-time physiotherapy instruction.

ELIGIBILITY:
Inclusion Criteria:

• Patients aged 60 years or above with displaced PHFs (Neer's definition) including 2-, 3-, or 4-part fractures after a low energy trauma will be recruited.

Prior to first visit in the outpatient clinic all patients with PHFs will be screened for eligibility based on initial radiographs and medical records by an experienced orthopaedic consultant (senior author SB) at Zealand University Hospital, Køge, Denmark. The senior author classifies fracture categories.

• Patients should be cognitively capable of answering patient-reported outcome measures.

Exclusion Criteria:

* Dependent on daily personal care for basic activities of daily living
* Diagnosed with dementia or institutionalized
* Does not understand written and spoken guidance in Danish
* Pathological fracture or previous fracture in the same proximal humerus
* Concomitant injury or fracture.
* Polytrauma, high-energy trauma, or multiple fractures
* Fracture dislocation or articular surface fracture
* Isolated tuberosity fracture
* Fractures not expected to heal by non-surgical treatment (no bony contact between head and shaft in both views)
* The senior author considers the patient unsuitable to attend the study for medical reasons (substance abuse, affective or psychotic disorders, apoplexy, chronic pain, malignant disease)
* Symptomatic glenohumeral osteoarthritis, rheumatoid arthritis, or rotator cuff-arthropathy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Oxford Shoulder Score (OSS) | 6 months
  Patient administered shoulder specific score, score ranges between between 0 and 48, with a higher score implying a greater degree of disability.

SECONDARY OUTCOMES:
European Quality of life-5 Dimensions-Three-Level (EQ-5D-3L) | 6 months
  Health-related quality of life, index score: < 0 to 1 (full health), with anchoring of death as 0.
European Quality of life-5 Dimensions-Three-Level (EQ-5D-3L) | 12 months
  Health-related quality of life, index score: < 0 to 1 (full health), with anchoring of death as 0.
Conversion to surgery | 6 months
  Number of patients converting to surgery
Oxford Shoulder Score (OSS) | 12 months
  Patient administered shoulder specific score, score ranges between between 0 and 48, with a higher score implying a greater degree of disability.

OTHER OUTCOMES:
European Quality of life-5 Dimensions-Three-Level (EQ-5D-3L) visual analogue scale | 6 months
  The patient's own health 'today' is rated between 0 (worst imaginable health) and 100 (best imaginable health)
European Quality of life-5 Dimensions-Three-Level (EQ-5D-3L) visual analogue scale | 12 months
  The patient's own health 'today' is rated between 0 (worst imaginable health) and 100 (best imaginable health)

CONTACTS AND LOCATIONS:
Overall Officials: Behnam Liaghat, MSc, Principal Investigator — Zealand University Hospital, University of Southern Denmark; Stig Brorson, PhD, Study Director — Zealand University Hospital, University of Copenhagen
Locations (1):
- Department of Orthopaedics, Zealand University Hospital, Køge, Denmark

IPD SHARING:
Plan to Share IPD: No
Anonymised data on group level will be made available upon reasonable request after the primary publications have been published.

REFERENCES:
- [Derived] Liaghat B, Brorson S. Effect of structured rehabilitation versus non-structured rehabilitation following non-surgical management of displaced proximal humerus fractures: a protocol for a randomised clinical trial. BMJ Open. 2022 Oct 17;12(10):e064156. doi: 10.1136/bmjopen-2022-064156. PMID 36253041